CLINICAL TRIAL: NCT02074696
Title: The Effect of BDNF on Motor Learning
Brief Title: BDNF and Motor Learning
Acronym: BDNF
Status: Terminated | Type: Observational
Why Stopped: Site unable to complete full data collection/protocol
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1401M46962
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: BDNF; Polymorphism, Genetic
Keywords: brain derived neurotrophic factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva sample for BDNF testing
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to assess the status of brain-derived neurotrophic factor brain (BDNF) and how the brain behaves in response to skill acquisition. Specifically we will investigate the relationship of the status of BDNF with cortical excitability changes and learning that occur during a motor training paradigm. We aim to 1) determine cortical excitability changes by using transcranial magnetic stimulation (TMS) before and after training; 2) to determine finger tracking accuracy before and after training; and 3) determine the presence of BDNF polymorphism in each participant.

We are testing healthy adults in this study, and eventually would like to apply to persons who have neurologic disorders such as stroke or dystonia. By applying a magnetic field to the outside of the head, electrical currents are produced within the brain that can stimulate brain tissue. Using TMS, the brain can be studied to gain a greater understanding of the mechanisms associated with cortical excitability in healthy and patient populations. There is limited knowledge of what influence genetic biomarkers such as BDNF have on cortical excitability changes within the cortex following learning. Studies have indicated that people without this certain gene are less likely to show changes in brain excitability during TMS and during motor learning than people with this gene

DETAILED DESCRIPTION:
Subjects and Design: A pretest/posttest design will be used. A convenience sample of healthy college students will be studied and will undergo an initial screening by the PI or Co-Investigators consisting of medical history and neurologic disorder review to assess safety and qualifications to participate.

Inclusion/ Exclusion Criteria: Inclusion criteria include ages between 18-45 years and no past history of psychiatric or neurologic disease. Exclusion criteria include subjects with any neuromuscular disorder that impairs upper extremity motion or seizure history. Subjects cannot be pregnant nor have indwelling metal or medical devices that are incompatible with TMS testing.

With the subject seated in a supportive chair, the subject's skin will be cleaned surrounding the first doral interoseus belly and dorsum of the hand. Next small surface electromyographic (EMG) electrodes will be attached at the muscle belly and tendon. A ground electrode will be placed on the dorsum of the hand or wrist.

Next, the threshold for TMS activation of the target muscle will be determined. To find the optimal position for activating the first dorsal interosseous muscle, we will use a 70-mm figure-eight TMS coil connected to a Magstim rapid magnetic stimulator. The coil will be handheld on the scalp over the approximate area of the primary motor cortex (M1) in the contralateral hemisphere to the recording electrode, and moved systematically to find the optimal position. Single-pulse magnetic stimuli will be delivered manually at approximately 0.1 Hz starting at an intensity of 50% of the stimulator maximum. This level will be adjusted systematically until the resting motor threshold is found, defined as the minimum intensity required to elicit a motor evoked potential (MEP) >50 µV peak-to-peak in at least 5 of 10 trials with the target muscle at rest. Various cortical excitability measures will be collected lasting approximately 20 minutes.

Finger tracking/training will be provided for 30 minutes under the supervision of the PI or Co-I. Subjects will wear a finger electrogoniometer at the index finger metacarpophalangeal (MP) joint. Subjects will use flexion/extension movements of the respective joint to track waveforms on a computer screen. The training would consist of 30 blocks of tracking trials. Each block will consist of 3 trials. The protocol parameters for different blocks will differ in waveform, amplitude, frequency, trial duration, and joint position. For example, a square wave would involve a different movement pattern execution as opposed to a triangular wave. The waveforms may also differ on the forearm position to create "stimulus-response compatible" or "stimulus-response incompatible" conditions. For example, a stimulus-response incompatible joint position would involve extending and flexing the joint (finger MP or elbow) in the horizontal plane to produce cursor movements in the vertical plane. All these factors challenge the individual's capabilities to problem solve to achieve optimum learning.

Following training and accuracy testing, cortical excitability measures will be collected again lasting approximately 20 minutes. Lastly, a saliva sample will be collected for genetic screening for brain derived neurotrophic factor (BDNF) polymorphism. We will collect approximately 2 ml (less than one-half teaspoon) of saliva by asking the subject to spit into a tube. It may take up to 30 minutes to provide a saliva sample, however, most people typically require less time (approximately 5 minutes).

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* no past history of psychiatric or neurologic disease.

Exclusion Criteria:

* any neuromuscular disorder that impairs upper extremity motion or seizure history
* Pregnancy
* Indwelling metal or medical device that are incompatible with TMS testing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Accuracy Index | Day 1: posttest after training
  A computer quantified tracking performance measure in each test. This is a calculation of accuracy by using the equation: AI = 100(P-E)/P. Where E is the root mean square (r.m.s.) error between the target line and the response line, and P is the size of the individual's target pattern, calculated as the r.m.s. difference between the sine wave and the midline separating the upper and lower phases of the sine wave. The magnitude of P is determined by the scale of the vertical axis, which is the subject's range of finger motion. Therefore, the AI is normalized to each subject's own range of motion and takes into account any differences between subjects in the excursion of the tracking target. The maximum possible score is 100%. Negative scores occur when the response line is so distant from the target that it falls on the opposite side of the midline.

SECONDARY OUTCOMES:
Cortical Excitability | Day 1: baseline
  Cortical excitability will be measured with transcranial magnetic stimulation (TMS) single and paired pulse stimulation to measure short-interval intracortical inhibition (SICI), cortical silent period (CSP) and motor evoked potential (MEP) amplitude.
Cortical Excitability | Day 1: posttest
  Cortical excitability will be measured with transcranial magnetic stimulation (TMS) single and paired pulse stimulation to measure short-interval intracortical inhibition (SICI), cortical silent period (CSP) and motor evoked potential (MEP) amplitude.

OTHER OUTCOMES:
BDNF genetic status | Day 1
  BDNF genetic variant screening will be conducted via saliva sample collected at the end of the session on day 1. We will screen for the Val66met polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J Kimberley, PhD, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States